CLINICAL TRIAL: NCT01230632
Title: Metabolic Phenotyping of Individuals Born Following Assisted Reproduction
Brief Title: Metabolic Phenotyping of Individuals Born Following Assisted Reproduction Techniques
Acronym: IMPART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Miaoxin Chen, Dr., University of Adelaide
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 100510a
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Syndrome; Diabetes
Keywords: assisted reproduction technology; Metabolic risk factors; In Vitro Fertilisation
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary Supplement (Experimental): 3 days high fat food
  Interventions: Dietary Supplement: high fat overfeeding

INTERVENTIONS:
Dietary Supplement: high fat overfeeding — Dietary Supplement:3 days overfeeding
  Other Names: 3 days overfeeding

SUMMARY:
This study is to compare the effects of high fat overfeeding on metabolic risk factors in children born though assisted reproduction technologies (ART) versus children conceived naturally (controls). The investigators will utilize state of the ART measures to characterize the physiological, endocrine and molecular responses to high fat overfeeding.

The investigators hypothesize that children conceived following ART will have greater responses to high fat dietary challenge and that this will be associated with DNA hypermethylation of genes that are involved in lipid metabolism.

DETAILED DESCRIPTION:
This study represents a novel initiative by the investigators to determine whether children conceived through ART have different metabolic responses at baseline or in response to high fat overfeeding as compared to age and body mass index-matched spontaneously conceived controls. Furthermore, the investigators will identify any differences in DNA methylation of candidate genes involved in lipid metabolism in adipose tissue and blood, to determine whether this is related to adverse outcomes during high fat overfeeding. The results from this study will help answer growing questions of the future health of In vitro fertilisation (IVF) babies, and may stimulate further research into optimising protocols for ovarian stimulation or in-vitro conditions during early blastocyst development.

ELIGIBILITY:
Inclusion Criteria:

* Post-pubertal healthy individuals aged 18-25years

Exclusion Criteria:

* Participants are ineligible if they have any significant medical conditions (e.g. personal history or clinical manifestation of cardiovascular disease, type 2 diabetes),
* strong family histories of diabetes or cardiovascular disease (e.g. first-degree relatives),
* take concomitant medications (eg: metformin),
* if they smoke or drink >140g of alcohol/week, , or
* were born prematurely (<37 weeks), or
* from mothers who had gestational diabetes.

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
intravenous glucose tolerance test (IVGTT) | 18 months
  After infusion of glucose bolus(0.3mg/kg, 50% glucose), blood samples are taken at 0,1,3,5,7,10,20,30 and 60 minutes. The value of glucose is recorded respectively (unit:mMol/L).

SECONDARY OUTCOMES:
insulin sensitivity | 18 months
  A 2-hour hyperinsulinemic euglycemic clamp (60mU/m2/min) is used to measure insulin sensitivity(µmol/min/kg Fat Free Mass). This is calculated by the formula from the amount of dextrose necessary to maintain blood glucose at 5mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Heilbronn, PhD, Principal Investigator — Department of Medicine
Locations (1):
- Leonie Heilbronn, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Chen M, Liu B, Wilkinson D, Hutchison AT, Thompson CH, Wittert GA, Heilbronn LK. Selenoprotein P is elevated in individuals with obesity, but is not independently associated with insulin resistance. Obes Res Clin Pract. 2017 Mar-Apr;11(2):227-232. doi: 10.1016/j.orcp.2016.07.004. Epub 2016 Aug 11. PMID 27524654
- [Derived] Chen M, Wu L, Zhao J, Wu F, Davies MJ, Wittert GA, Norman RJ, Robker RL, Heilbronn LK. Altered glucose metabolism in mouse and humans conceived by IVF. Diabetes. 2014 Oct;63(10):3189-98. doi: 10.2337/db14-0103. Epub 2014 Apr 23. PMID 24760136